CLINICAL TRIAL: NCT02676661
Title: The Prevalence and Risk Factors for Patients With Peri-implant Disease： A Prospective Study
Brief Title: Evaluation of the Prevalence and Risk Factors for Patients With Peri-implant Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Ji-hua Chen, Professor and Dean of the Department of Prosthodontics, School of Stomatology, Fourth Military Medical University, Air Force Military Medical University, China
Other Study IDs: Jhchen
Record Dates: First submitted 2016-01-24; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Jaw, Edentulous, Partially
Keywords: peri-implant disease; risk factors; prevalence
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- no peri-implant disease: The subjects who did not suffer from peri-implant disease.
- peri-implant disease: The subjects who suffered from peri-implant disease.

SUMMARY:
To investigate the prevalence and risk factors for peri-implant disease in partially edentulous patients rehabilitated with implants supported crown or bridge so as to provide evidence for clinical prevention and control.

DETAILED DESCRIPTION:
The aim of the present study is to identify the prevalence of peri-implant disease in partially edentulous subjects treated with osseointegrated implants, using clinical parameters, as well as to analyse the possible disease association with demographic, behavioural, and biological risk variables.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients will implant at least one implant and will be restored with implant-supported fixed partial dentures and single crowns.

Exclusion Criteria:

* Jaw radiotherapy treatment before and after implanting. Patients who have bruxism,xerostomia or the adjacent teeth periapical periodontitis.
* Patients who suffered with oral mucosa disease,or aggressive periodontitis or jaw defect.
* Patients who suffered with mental and psychological disease will influence their oral health normal maintenance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Partially edentulous patients implant dental implants and will be restored with implant-supported fixed partial dentures and single crowns at the Department of Prosthodontics, School of Stomatology of the Fourth Military Medical University
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2014-10; Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
peri-implant disease | at the 5 years after prosthetic loading.
  Peri-implant disease includes Peri-implant mucositis and Peri-implantitis.Peri-implant mucositis: BoP/suppuration but no detectable bone loss. Peri-implantitis: BoP/suppuration and bone loss >2 mm.

SECONDARY OUTCOMES:
Gingival Bleeding on Probing | at the first day,6 months 1,3 and 5 years after prosthetic loading.
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding.
Pocket depths | at the first day,6 months 1,3 and 5 years after prosthetic loading.
  PD will be measured from the free gingival margin to the base of the pocket and will be recorded in whole millimeters (mm).
Marginal bone loss | at the first day,6 months 1,3 and 5 years after prosthetic loading.
  Marginal bone loss will be assessed by periapical radiographs taken with the paralleling technique.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjin Chen, PhD, Principal Investigator — IRB of Stomatological Hospital of FMMU,PLA
Locations (1):
- Stomatological Hospital of Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes